CLINICAL TRIAL: NCT05580939
Title: The Effect of a Web-based Simulation Application Developed for Use in Basic Life Support Education on Nursing Students' Knowledge, Satisfaction and Self-Confidence Levels
Brief Title: The Effect of a Web-based Simulation Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Selin Keskin Kızıltepe, PhD, Duzce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DuzceUselin
Record Dates: First submitted 2022-10-08; First posted 2022-10-14 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Self Confidence; Knowledge, Attitudes, Practice; Satisfaction
Keywords: Basic life support; Web based simulation
MeSH Terms: conditions — Behavior; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: The study was conducted with a mixed-method design. In this study, there are two groups as intervention group and control group. Investigator, administered not any application to control group. Intervention group will use the web-based simulation application for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Grup (No Intervention): they receive theoretical first aid training
- Intervention Grup (Experimental): they receive theoretical first aid training and use web based simulation application
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: Intervention group — They use Web-based Simulation Application for 4 weeks
  Arms: Intervention Grup

SUMMARY:
Cardiopulmonary resuscitation (CPR) training for nursing students is important. The importance of using computer-assisted simulation in gaining skills for basic life support applications is increasing. In addition to the use of simulation-based teaching methods in many different fields, it is seen that they are also used for the development of cardiopulmonary resuscitation practices of students and produce effective results.The aim of the study is to evaluate the effect of a web-based simulation application used in basic life support education on the level of knowledge, satisfaction and self-confidence of nursing students.

DETAILED DESCRIPTION:
This research was conducted with 60 nursing student (intervention group: 30, control group: 30). The study is a mixed method type randomized controlled intervention study in which quantitative and qualitative research methods are used together.The quantitative data were obtained by using the ""Basic Life Support Knowledge Form", "Basic Life Support Skill Form", "Student Satisfaction and Self Confidence in Learning Scale, Perceived Learning Scale" , and the qualitative data were collected by using the "Semistructured Interview Form" in focus group sessions.

ELIGIBILITY:
Inclusion Criteria:

Being nursing student

Exclusion Criteria:

no previous training in basic life support not filling out the questionnaires completely

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Basic life support level of knowledge and skill | post-test will be administered four weeks later (pre-test will be performed in the first week)
  Data were collected via " basic life support knowledge and skill scale". The minimum score taken from the scale is 0 and the maximum score is 20. Higher score indicate that there is a high level of knowledge and skill.Students using a web-based simulation application have higher knowledge and skill.
level of self confidence | post-test will be administered four weeks later (pre-test will be performed in the first week)
  Data were collected via " Student Satisfaction and Self-Confidence in Learning Scale ". The minimum score taken from the scale is 13 and the maximum score is 65. Higher score indicate that there is a high level of self confidence. Students using a web-based simulation application have higher self-confidence score than other students.
level of satisfaction | post-test will be administered four weeks later (pre-test will be performed in the first week)
  Data were collected via " Student Satisfaction and Self-Confidence in Learning Scale ". The minimum score taken from the scale is 13 and the maximum score is 65. Higher score indicate that there is a high level of satisfaction.Students using a web-based simulation application have higher satisfaction score than others

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Suarez M, Mendez-Martinez C, Martinez-Isasi S, Gomez-Salgado J, Fernandez-Garcia D. Basic Life Support Training Methods for Health Science Students: A Systematic Review. Int J Environ Res Public Health. 2019 Mar 3;16(5):768. doi: 10.3390/ijerph16050768. PMID 30832440
- [Background] Boada I, Rodriguez-Benitez A, Garcia-Gonzalez JM, Olivet J, Carreras V, Sbert M. Using a serious game to complement CPR instruction in a nurse faculty. Comput Methods Programs Biomed. 2015 Nov;122(2):282-91. doi: 10.1016/j.cmpb.2015.08.006. Epub 2015 Aug 21. PMID 26319184